CLINICAL TRIAL: NCT02526680
Title: The Impact of a Novel Artificial Vision Device (OrCam) on the Quality of Life of Patients With Advanced Glaucoma
Brief Title: Does Using a Low Vision Aid Device Improve Quality of Life in Glaucoma Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-396
Record Dates: First submitted 2015-08-06; First posted 2015-08-18 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma
Keywords: OrCam; Low-vision device; End-stage glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Glaucoma Subjects (Experimental): 27 glaucoma subjects will be given the OrCam low vision aid device to use for 1 month.
  Interventions: Device: OrCam

INTERVENTIONS:
Device: OrCam — The OrCam low vision aid, camera attached to glasses, used by 27 glaucoma subjects for 1 month.

SUMMARY:
To determine the impact of OrCam over 1 month on health-related quality of life (HRQoL) in subjects with advanced glaucoma using the National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ-25).

To identify tasks for which subjects are using the OrCam device and patient satisfaction.

DETAILED DESCRIPTION:
Participants will document their daily impression about the use of OrCam, a small camera attached to their glasses over a 1-month period. They will attend 2 appointments at Wills Eye Hospital Glaucoma Research Center (baseline and final visit). Participant's will be trained to use the OrCam device at baseline visit and complete a best-corrected visual acuity assessment ETDRS (early treatment diabetic retinopathy study) and the NEI-VFQ-25 questionnaire. They will also read a short newspaper article.

The NEI-VFQ-25 includes a series of 25 questions pertaining to vision or feelings about a vision condition. Answers are selected among a numbered list of possible responses, the values of which are ultimately recoded and converted to a 0 to 100 scale. Items within each subscale are averaged together to create 12 subscale scores. An overall composite score will be calculated by averaging vision-targeted subscale scores, excluding the general health rating question.

Participants will read a short article. They will be asked to grade their reading difficulty between 1 (unable to read) to 10 (able to read without difficulty). Time to read article will be recorded. Reading task will be performed with best correction - with and without the assistance of the OrCam device.

Subjects will utilize OrCam daily for one month. Each week, subjects will record thoughts about the device in a log book or by using audio tape recorder, according to patient's personal preference.

Final assessment at 1 month will include best-corrected visual acuity (ETDRS), NEI-VFQ-25, and the newspaper-reading task with and without OrCam assistance. A satisfaction questionnaire will be completed in order to assess subjects' overall feelings regarding OrCam. Audio log books will be analyzed for specific factors and recorded by a research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma any type, characterized by glaucomatous optic neuropathy and corresponding visual field (VF) defect
* Visual acuity of 20/400 to hand motion (HM) in better eye or visual field less than 10 degrees in better eye and having difficulty reading.
* Age 18 years or older
* Able to understand and speak English
* Able to use an electronic recording device
* Able to operate a computerized system

Exclusion Criteria:

* Neurological or musculoskeletal problems that would influence performance on activities of daily living
* Incisional eye surgery within past three months
* Laser therapy within previous month
* Any cause for visual impairment other than glaucoma
* Photophobia
* Any medical condition precluding subject from providing reliable, valid data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Jay Katz, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Manuscript accepted for publication August 2018.

RESULTS

PARTICIPANT FLOW:
Groups:
- Glaucoma Subjects: 27 glaucoma subjects were given the OrCam low vision aid device to use for one month. National Eye Institute Visual Function Questionnaire - 25 (NEI-VFQ-25) was administered at baseline and 1 month.
Period: Overall Study
Arm/Group | Glaucoma Subjects
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [22 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Impact of OrCam on Vision-related Quality of Life
Description: National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) is a series of questions pertaining to vision or feelings about a vision condition in relation to functional status to assess their quality of life. Multiple choice responses from 12 subscales (general vision, near vision, distance vision, ocular pain, social functioning, mental health, roll difficulties, dependency, driving, color vision and peripheral vision) were recorded into a 0-100 score where 0 represents the lowest perceived vision difficulties and 100 the highest perceived difficulties. NEI-VFQ-25 was used to measure the number of participants who showed improvement in vision-related quality of life after using the OrCam device over a one month period.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Glaucoma Subjects: 27 glaucoma subjects were given the OrCam low vision aid device to use for one month. National Eye Institute Visual Function Questionnaire - 25 (NEI-VFQ-25) was administered at baseline and 1 month after using the device to measure improvement in perceived vision-related quality of life.
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 27
Participants | 20

2. Secondary Outcome: Impact of OrCam on Reading Newspapers
Description: Participants were asked 'Did OrCam increase your quality of life in reading newspapers?' after a one month trial period with the device. Number of subjects answering Yes is provided.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Glaucoma Subjects: 27 glaucoma subjects were given the OrCam low vision aid device to use for 1 month.
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 27
Participants | 15

3. Secondary Outcome: Impact of OrCam on Grocery Shopping
Description: Participants were asked 'Did OrCam improve your quality of life while grocery shopping?' after a one month trial period with the device. Number of subjects answering Yes is provided.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 27
Participants | 5

4. Secondary Outcome: Recommending OrCam to Others
Description: Participants were asked 'How likely would you be to recommend OrCam to another visually impaired person?' after a one month trial period with the device. Number of subjects answering Very Likely or Likely is provided.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 27
Participants | 23

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Glaucoma Subjects
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
OrCam device requires further improvement. Cost of OrCam poses limitation on access to many individuals and is not covered by most health insurance plans in the United States for visually impaired patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No